CLINICAL TRIAL: NCT07393698
Title: Effectiveness of a Personalized Online Intervention for Optimizing Time Allocation Across 24-hour Movement Behaviours in College Students: a Randomized Controlled Trial
Brief Title: Intervention to Improve 24-Hour Movement Behaviors in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South China Normal University (Other)
Responsible Party: Principal Investigator, Ru ZHANG, Associate Professor; Principal Investigator, South China Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SCNU-SPT-2023-175; 22YJC890050 (Other Grant/Funding Number: Ministry of Education of China)
Record Dates: First submitted 2026-01-16; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Physical Activity; Sedentary Behaviour; Sleep
Keywords: time allocation; 24-hour movement behaviour
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention group: Personalized one-on-one guidance was delivered via WeChat twice weekly, with each session lasting approximately 15 minutes. Guidance content was individualized based on participants' baseline 24-hour movement behaviour profiles, with the explicit aim of promoting more optimal time-use patterns across daily behaviours. In addition, participants were invited to attend weekly, 30-minute offline group jogging sessions, during which heart rate was maintained within individually prescribed target ranges. The participants were encouraged to achieve behavior goals. Participants allocated to the control group received no intervention during the study period and were asked to maintain their usual lifestyle and daily routines.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the personalized online intervention, participants and intervention providers were not blinded to group allocation. Outcome assessors were blinded to group assignment, and participants were instructed not to disclose their allocation status during outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 24-hour Movement Behaviour Intervention (Experimental): Personalized one-on-one guidance was delivered via WeChat twice weekly, with each session lasting approximately 15 minutes. Guidance content was individualized based on participants' baseline 24-hour movement behaviour profiles, with the explicit aim of promoting more optimal time-use patterns across daily behaviours. In addition, participants were invited to attend weekly, 30-minute offline group jogging sessions, during which heart rate was maintained within individually prescribed target ranges. Participants were encouraged to achieve behaviour goals.
  Interventions: Behavioral: Personalized Online Behavioral Intervention
- Usual Practice Control (No Intervention): Participants allocated to the control group received no intervention during the study period and were asked to maintain their usual lifestyle and daily routines. They did not receive personalized guidance, structured PA sessions, behavioural monitoring, or incentives

INTERVENTIONS:
Behavioral: Personalized Online Behavioral Intervention — The intervention consisted of a personalized, online behavioural program delivered via WeChat, in order to support more optimal allocation of daily time across physical activity, sedentary behaviour, and sleep within a finite 24-hour day. Intervention content was individualized based on each participant's baseline 24-hour movement behaviour profile. Personalized feedback and guidance were based on the Multi-Process Action Control (M-PAC) framework. participants in the intervention group were invited to attend weekly 30-minute offline group jogging sessions.
  Arms: 24-hour Movement Behaviour Intervention

SUMMARY:
This study examined whether a personalized, WeChat-based behavioural intervention could help improve how university students allocate their time across daily movement behaviours, including physical activity, sedentary behaviour, and sleep.

University students were randomly assigned to either an intervention group or a control group. Participants in the intervention group received individualized guidance, feedback, and behaviour-change support delivered through WeChat. The intervention was designed to help participants develop more balanced daily movement behaviour patterns within a 24-hour day. Participants in the control group continued their usual routines without receiving intervention materials.

The primary outcome of the study was the time-use composition of 24-hour movement behaviours, reflecting how daily time was distributed across physical activity, sedentary behaviour, and sleep. Psychological factors related to behaviour regulation, such as motivation, planning, and habit, were also assessed.

The results of this study aim to inform the development of theory-informed, personalized digital interventions that support healthier daily movement behaviour patterns among university students.

DETAILED DESCRIPTION:
This randomized controlled behavioural study was conducted to evaluate the effectiveness of a personalized, online intervention based on the Multi-Process Action Control (M-PAC) framework in optimizing the time-use composition of 24-hour movement behaviours among university students.

Participants were randomly assigned to either an intervention group or a control group. The intervention group received a personalized behavioural program delivered via WeChat. The program was designed to support more optimal allocation of daily time across physical activity, sedentary behaviour, and sleep by targeting key behavioural processes, including reflective, regulatory, and reflexive mechanisms. Intervention content included individualized feedback and behaviour-change support tailored to each participant's movement behaviour profile. The control group did not receive intervention materials and continued their usual daily routines.

The primary outcome was the time-use composition of 24-hour movement behaviours, defined as the relative distribution of time allocated to physical activity, sedentary behaviour, and sleep within a finite 24-hour period. Secondary outcomes comprised psychological constructs related to behaviour regulation, derived from the Multi-Process Action Control (M-PAC) framework. These constructs included affective attitude, instrumental attitude, perceived capability, perceived opportunity, intention, planning, self-monitoring, identity, and habit, and were assessed using validated Chinese-language self-report questionnaires with established psychometric properties. In the present study, healthy time allocation of 24-hour movement behaviours was operationally defined in accordance with the Canadian 24-Hour Movement Guidelines for Adults, which recommend regular engagement in moderate-to-vigorous physical activity, participation in light-intensity physical activity across the day, limited recreational screen time, adequate sleep duration, and regular muscle-strengthening activities.

The study involved a non-clinical population and did not include biomedical or medical health outcomes. The study protocol was approved by the institutional ethics committee, and written informed consent was obtained from all participants prior to participation.

ELIGIBILITY:
Inclusion Criteria

1. aged 18-25 years;
2. no severe physical or psychological conditions, no contraindications to exercise, and no major surgery in the past six months;
3. willingness to wear an accelerometer and participate in the online intervention;
4. failure to meet at least one recommendation of the Canadian 24-Hour Movement Guidelines for Adults (18-64 years) for PA, sedentary behaviour, or sleep -

Exclusion Criteria:

1. Presence of severe physical or psychological conditions that could limit safe participation in physical activity.
2. Medical contraindications to exercise or a history of major surgery within the past six months.
3. Inability or unwillingness to wear an accelerometer or to engage in the online intervention.
4. Meeting all recommendations of the Canadian 24-Hour Movement Guidelines for Adults (18-64 years) at baseline.

   -

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Time allocation of 24-hour movement behaviour | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Time allocation of 24-hour movement behaviours was objectively assessed using a waist-worn ActiGraph GT3X accelerometer worn continuously for seven consecutive days.

SECONDARY OUTCOMES:
Affective attitude toward healthy 24-hour movement behaviour time allocation (Theory of Planned Behaviour Questionnaire) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Affective attitude toward healthy time allocation of 24-hour movement behaviours was assessed using three bipolar adjective pairs (unpleasant-pleasant, boring-interesting, and unenjoyable-enjoyable) adapted from established Theory of Planned Behaviour questionnaires (https://people.umass.edu/aizen/pdf/tpb.measurement.pdf). Participants responded to a common stem ("In the next week, compliance with healthy time allocation of 24-hour movement behaviours is …"), followed by three items. Responses were recorded on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). A mean score was calculated across the three items, with higher scores indicating a more positive affective attitude.
Instrumental attitude toward Healthy 24-Hour Movement Behaviour Time Allocation (Theory of Planned Behaviour Questionnaire) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Instrumental attitude was assessed using three bipolar adjective pairs (harmful-beneficial, worthless-valuable, and bad-good) adapted from established Theory of Planned Behaviour measures (https://people.umass.edu/aizen/pdf/tpb.measurement.pdf
  ). Participants responded to a common stem ("In the next week, compliance with healthy time allocation of 24-hour movement behaviours is …"), followed by three items (e.g., "In the next week, compliance with healthy time allocation of 24-hour movement behaviours is harmful-beneficial"). Responses were recorded on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). A mean score was calculated across the three items, with higher scores indicating a more positive instrumental attitude.
Perceived capability toward healthy 24-hour movement behaviour time allocation (Theory of Planned Behaviour Questionnaire) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Perceived capability was assessed using three items adapted from established Theory of Planned Behaviour measures (https://people.umass.edu/aizen/pdf/tpb.measurement.pdf
  ). Participants responded to a common stem ("In the next week, compliance with healthy time allocation of 24-hour movement behaviours is …"), followed by items assessing perceived ease and capability (e.g., "It is easy for me to comply with healthy time allocation of 24-hour movement behaviours in the next week"). Responses were recorded on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). A mean score was calculated across the three items, with higher scores indicating greater perceived capability.
intention toward healthy 24-hour movement behaviour time allocation (Theory of Planned Behaviour Questionnaire) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Intention was assessed using three items adapted from established Theory of Planned Behaviour measures (https://people.umass.edu/aizen/pdf/tpb.measurement.pdf
  ). Participants responded to a common stem ("In the next week, compliance with healthy time allocation of 24-hour movement behaviours is …"), followed by items assessing behavioural intention (e.g., "I intend to comply with healthy time allocation of 24-hour movement behaviours in the next week"). Responses were recorded on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree). A mean score was calculated across the three items, with higher scores indicating stronger intention.
Perceived opportunity toward healthy 24-hour movement behaviour time allocation (Multi-Process Action Control Questionnaire) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Perceived opportunity was assessed using three items adapted from the questionnaire based on the Multi-Process Action Control framework applied to individual physical activity. Items assessed participants' perceived opportunity to comply with healthy time allocation of 24-hour movement behaviours over the subsequent week (e.g., "If I really wanted to comply with healthy time allocation of 24-hour movement behaviours over the next week, I would have the opportunity to do so"). Responses were recorded on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). A mean score was calculated across the three items, with higher scores indicating greater perceived opportunity.
Planning towards healthy 24-hour movement behaviour time allocation (Health Action Process Approach Questionnaire) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Planning was assessed using six items adapted from questionnaires based on the Health Action Process Approach. Items assessed participants' use of planning strategies related to compliance with healthy time allocation of 24-hour movement behaviours over the previous week (e.g., "I made regular plans concerning how to comply with healthy time allocation of 24-hour movement behaviours in the last week"). Responses were recorded on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). A mean score was calculated across the six items, with higher scores indicating greater use of planning strategies.
Self-monitoring toward healthy 24-hour movement behaviour time allocation (Multi-Process Action Control Questionnaire) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Self-monitoring was assessed using three items adapted from questionnaires based on the Health Action Process Approach. Items assessed participants' engagement in monitoring their time allocation of 24-hour movement behaviours over the previous week (e.g., "I kept track of my time allocation of 24-hour movement behaviours in a diary or log over the last week"). Responses were recorded on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). A mean score was calculated across the three items, with higher scores indicating greater use of self-monitoring strategies.
Identity towards healthy 24-Hour movement behaviour time allocation (Exercise Identity Scale) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Identity was assessed using four items adapted from the Exercise Identity Scale. Items assessed the extent to which engagement in healthy time allocation of 24-hour movement behaviours was integrated into participants' self-concept (e.g., "When I describe myself to others, I usually include my involvement in healthy time allocation of 24-hour movement behaviours"). Responses were recorded on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). A mean score was calculated across the four items, with higher scores indicating stronger identity integration.
Habit towards healthy 24-hour movement behaviour time allocation (Self-Report Habit Index) | Baseline, Week 8 (post-intervention), and Week 16 (follow-up)
  Habit strength was assessed using twelve items adapted from the Self-Report Habit Index. Participants responded to a common stem ("In the last month, compliance with healthy time allocation of 24-hour movement behaviours was …"), followed by items assessing behavioural automaticity and repetition (e.g., "… something I do frequently"). Responses were recorded on a 5-point Likert scale (1 = strongly disagree, 5 = strongly agree). A mean score was calculated across the twelve items, with higher scores indicating stronger habit strength.

CONTACTS AND LOCATIONS:
Overall Officials: Ru ZHANG, Principal Investigator — South China Normal University
Locations (1):
- School of Physical Education and Sports Science, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No